CLINICAL TRIAL: NCT02544646
Title: Changes in Ocular Rigidity After Trabeculectomy in Patients With POAG or PEX
Brief Title: Changes in Ocular Rigidity After Trabeculectomy in Patients With POAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc.Prof. Priv.-Doz. MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-040411
Record Dates: First submitted 2014-02-19; First posted 2015-09-09 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma
Keywords: trabeculectomy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Exfoliation Syndrome

ARMS (1):
- trabeculectomy (Other)
  Interventions: Other: Changes in Ocular rigidity

INTERVENTIONS:
Other: Changes in Ocular rigidity — measured before the operation and 28±7 days after the operation

SUMMARY:
It has been hypothesized that the biomechanical properties of the optic nerve head and/or sclera play a role in the development of glaucoma. One approach of gaining insight into the biomechanical properties of the eye by the means of clinical studies is based on the Friedenwald equation, representing a pressure-volume relationship. This equation represents the so called ocular rigidity, which expresses the elasticity of the globe.

In order to be able to solve the equation, measurements of fundus pulsation amplitude (FPA) with laser interferometry and dynamic contour tonometric assessment of the pulse amplitude (PA) have to be performed.

In addition choroidal thickness will be assessed with OCT before and after trabeculectomy, since results in choroidal thickness measurements in patients with glaucoma are controversial.

The focus of this study lies on the changes of ocular rigidity and choroidal thickness after surgical trabeculectomy in patients with primary open angle glaucoma (POAG) or pseudoexfoliation glaucoma (PEX).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Normal ophthalmic findings except POAG or Pseudoexfoliation glaucoma (PEX)
* Patients scheduled for trabeculectomy

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceeding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Other types of glaucoma, such as pigmentary glaucoma, history of acute angle closure
* History of previous glaucoma surgery
* Postoperative IOP ≤ 8 mmHg
* Ocular inflammation or infection within the past 3 months
* Topical treatment with any ophthalmic drug except anti-glaucomatous medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Change in ocular rigidity | Baseline and 28±7 days postoperative
  Change in ocular rigidity after surgery

SECONDARY OUTCOMES:
Fundus pulsation amplitude | Baseline and 28±7 days postoperative
Ocular pulse amplitude | Baseline and 28±7 days postoperative
Mean arterial pressure | Baseline and 28±7 days postoperative
Pulse rate | Baseline and 28±7 days postoperative
Axial eye length | Baseline and 28±7 days postoperative
choroidal thickness | Baseline and 28±7 days postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria